CLINICAL TRIAL: NCT03637842
Title: Randomized Controlled Trial of Lorcaserin for Cannabis Use Disorder
Brief Title: Lorcaserin for Cannabis Use Disorder
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: terminated due to lorcaserin recall
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Christina Ann Brezing, Clinical Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7662
Record Dates: First submitted 2018-07-19; First posted 2018-08-20 (Actual); Results first posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Cannabis Use Disorder
Keywords: cannabis; impulsivity
MeSH Terms: conditions — Marijuana Abuse; Impulsive Behavior | interventions — lorcaserin

STUDY DESIGN:
Intervention Model Description: Double Blind Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Encapsulated medication
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lorcaserin XR (Active Comparator): Lorcaserin XR 20mg daily
  Interventions: Drug: Lorcaserin
- Placebo (Placebo Comparator): Placebo Oral Capsule
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Lorcaserin — Lorcaserin XR 20mg per day
  Other Names: Belviq
  Arms: Lorcaserin XR
Drug: Placebo oral capsule — Placebo
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to investigate the effect of lorcaserin on reductions in cannabis use and multiple constructs of impulsivity in outpatient treatment-seeking individuals with cannabis use disorder (CUD). Additionally, the investigators will make use of the technological application of ecological momentary assessments (EMA), to collect real-time data at key time intervals during the study on participants' use of cannabis and other substances in addition to measuring impulsive traits through self-initiated, fixed and random phone prompts. This will be a 13-week randomized, double-blind, placebo-controlled trial, with week 1 focused on baseline assessments of impulsivity (through EMA in vivo and at study visits), weeks 2- 3 of medication lead-in, and week 4 targeting a reduced cannabis use/quit day through week 13. The primary aims are to (1) Examine the effect of lorcaserin compared to placebo, on reductions in cannabis use among treatment-seeking outpatients with CUD, (2) Examine the effect of lorcaserin compared to placebo on behavioral and self-report measures of impulsivity among individuals with CUD during the medication lead-in phase (weeks 2-3). The secondary aim is to examine whether reductions in impulsivity (during weeks 2-3) mediates the effect of lorcaserin on cannabis use (during weeks 8-13), if the primary hypotheses are supported. Finally, the investigators will explore the effect of lorcaserin compared to placebo on (1) drop-out rates, (2) time to discontinuation from study, (3) treatment adherence, and (4) nicotine use.

DETAILED DESCRIPTION:
Cannabis use disorder (CUD) is a major public health problem associated with significant psychiatric and medical morbidity, poor performance, and legal consequences.4 4.2 million people in the United States meet criteria for CUD.5 15% of all admissions for substance abuse treatment were related to cannabis as the primary, presenting problem in 2014 and 86% of those admissions were referred for ambulatory care.6 Despite the large number of patients with CUD seeking outpatient treatment, the investigators have limited options available. While evidence-based practices (EBP), and specifically psychotherapies, have been studied to treat CUD and various approaches have been shown to have clinical utility,7-9 many patients have difficulty achieving significant reductions in their use or sustained abstinence.10 This is further complicated by patients' limited access to EBPs,11 frequent poor adherence by therapists in the community to EBP interventions,12-14 and challenges in treating CUD with EBPs when available in community settings.10 Finding effective medications for the treatment of CUD is essential. There are no FDA approved medications for CUD. A number of pharmacological treatment trials for CUD have been performed.1* While some agents have shown promise,15-17 no medication strategy has emerged as clearly efficacious in producing abstinence.1,18 As the changing legal landscape influences patients' goals for reductions in cannabis use as compared to abstinence only, and with increasing support from the research community, future studies need to identify medications that lead to reductions in cannabis use.

Impulsivity has been linked to the predisposition,19 severity,20 and poor treatment outcomes21, 22 in cannabis users and CUD, making it a prime pharmacology target. Notably, there is an entwined relationship between cannabis and impulsivity. Impulsivity as a neurobehavioral trait is associated with cannabis use,and acute and chronic use of cannabis has been shown to exacerbate impulsivity, with some mixed evidence likely attributable to diverse constructs of impulsivity used across studies. While the investigators may not be able to fully determine which came first-the impulsivity or the cannabis use, further research is needed to demonstrate whether reductions across constructs of impulsivity can lead to improvements in CUD, and vice versa. Over the last two decades, 5HT2C receptor agonists have been shown to alter neurobiological systems of addiction and relevant drug use behavior in the preclinical literature by increasing inhibitory control on mesolimibic dopamine processes and resultant incentive motivation based behaviors,23 both directly and indirectly, particularly with regards to their impact on reducing impulsivity.24 In 2012, lorcaserin, a selective 5HT2C receptor agonist, was approved by the FDA, allowing for clinical exploration of its role in the treatment of substance use disorders, including CUD.25 Recently, a fully powered clinical trial of lorcaserin for tobacco smoking cessation was positive.26 The primary purpose of this study is therefore to investigate the effect of lorcaserin on reductions in cannabis use and multiple constructs of impulsivity in outpatient treatment-seeking individuals with CUD.

Additionally, the investigators will make use of the technological application of ecological momentary assessments (EMA), to collect real-time data at key time intervals during the study on participants' use of cannabis and other substances in addition to measuring impulsive traits through self-initiated, fixed and random phone prompts. This will be a 13-week randomized, double-blind, placebo-controlled trial, with week 1 focused on baseline assessments of impulsivity (through EMA in vivo and at study visits), weeks 2-3 of medication lead-in, and week 4 targeting a reduced cannabis use/quit day through week 13. This "proof of concept" study will provide Dr. Brezing with training in randomized controlled trial operations, multiple constructs to measure impulsivity, utilization of technology as a measurement tool, and identification of outcomes that may prove important to reductions in cannabis use.

Primary Aims:

(Aim 1) Examine the effect of lorcaserin compared to placebo, on reductions in cannabis use among treatment-seeking outpatients with CUD, with the primary outcome measured by average weekly mean episodes of any cannabis use (including edibles, vaping, and other variable potency cannabinoid products) per day. (Aim 2) Examine the effect of lorcaserin compared to placebo on behavioral and self-report measures of impulsivity among individuals with CUD during the medication lead-in phase (weeks 2-3).

Secondary Aim: If the hypotheses of the Primary Aims are supported, the investigators will examine whether reductions in impulsivity (during weeks 2-3) mediates the effect of lorcaserin on cannabis use (during weeks 8-13).

Exploratory Aims: To explore the effect of lorcaserin compared to placebo on (1) drop-out rates, (2) time to discontinuation from study, (3) treatment adherence, and (4) nicotine use.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals between the ages of 18-70
2. Meets DSM-V criteria for a current cannabis use disorder
3. Seeking treatment for cannabis use disorder
4. THC-positive urine drug screen
5. Capable of giving informed consent and complying with study procedures
6. Has regular access to the internet by any means
7. Not underweight (Defined as BMI ≥18.5)

Exclusion Criteria:

1. Lifetime history of DSM-V diagnosis of schizophrenia or schizoaffective disorder
2. Current DSM-V criteria for a psychiatric disorder supported by the MINI that in the investigator's judgment is unstable, would be disrupted by the study medication, or is likely to require new pharmacotherapy or psychotherapy during the study period. Individuals who are currently stable on psychotropic medication for at least 3months may be included if in the investigator's opinion the psychotropic medication is compatible with the study medication (lorcaserin).
3. Individuals who meet DSM-V criteria for any moderate to severe substance use disorder other an cannabis, caffeine or nicotine use disorders
4. Pregnancy, lactation, or failure to use adequate contraceptive method in female patients who are currently engaging in sexual activity with men
5. Unstable medical conditions, such as AIDS, cancer, uncontrolled hypertension, uncontrolled diabetes, pulmonary hypertension or heart disease; or individuals with a history of serotonin syndrome
6. Legally mandated to participate in a substance use disorder treatment program
7. Current or recent history of significant violent or suicidal behavior, risk for suicide or homicide
8. Currently meets DSM-V diagnosis for an eating disorder or is underweight (BMI <18.5)
9. Elevated liver function tests (AST and ALT > 3 times the upper limit of normal) or impaired renal function
10. Known history of allergy, intolerance, or hypersensitivity to lorcaserin
11. Concurrent use of migraine medications ergotamine (Cafergot, Ergomar) or dihydroergotamine (Migranal), 5HT2B receptor agonists like cabergoline, medications metabolized by CYP2D6 (thioridazine, tamoxifen, metoprolol, aripiprazole, codeine,, MAOIs, or St. John's Wort

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Brezing, MD, Principal Investigator — CUMC/NYSPI
Locations (1):
- Columbia Substance Treatment and Research Service, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 person who was enrolled dropped out of the study prior to randomization. 4 people were randomized in total.
Period: Overall Study
Arm/Group | Lorcaserin XR | Placebo
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lorcaserin XR | Placebo | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.0 (1.4) | 33.5 (16.3) | 28.8 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved a Reduction in Cannabis Use Per Daily Quartiles
Description: descriptive of cannabis use per day captured in daily quartiles based on self report as collected by the Time Line Follow back. The quartiles defined as follows: 12AM-6AM; 6AM-12PM; 12PM-6PM;6PM-12AM. Participants would report if they used during each of these times.
Time Frame: 13 weeks of study or participants length of participation
Measure: Number; unit: participants
Arm/Group | Lorcaserin XR | Placebo
Number analyzed (Participants) | 2 | 2
participants | 2 | 0

ADVERSE EVENTS:
Time Frame: Up to 13 weeks
Arm/Group | Lorcaserin XR | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
Study was prematurely terminated due to FDA recall of Lorcaserin.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/42/NCT03637842/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/42/NCT03637842/SAP_001.pdf